CLINICAL TRIAL: NCT05588193
Title: ED2PrEP - Patient Focused, Low-burden Strategies for PrEP Uptake Among Emergency Departments Patients: a Two-arm Hybrid Implementation-effectiveness Trial
Brief Title: ED2PrEP - Patient Focused, Low-burden Strategies for PrEP Uptake Among Emergency Departments
Acronym: ED2PrEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-13724; R01AI169636 (NIH)
Record Dates: First submitted 2022-10-07; First posted 2022-10-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: HIV

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post Visit Outreach (PVO) (Experimental): Outreach by trained patient navigators/educators after patients' ED visit for education, counseling, linkage to preventive/sexual health care.
  Interventions: Behavioral: PVO
- Tele-Sexual Healthcare (TSH) visit during the ED visit (Experimental): Tele-sexual health visit with a specialist offered during the ED visit to patients.
  Interventions: Behavioral: TSH

INTERVENTIONS:
Behavioral: PVO — post-visit outreach
  Arms: Post Visit Outreach (PVO)
Behavioral: TSH — tele-sexual health visit during the ED visit
  Arms: Tele-Sexual Healthcare (TSH) visit during the ED visit

SUMMARY:
Severe inequities in HIV pre-exposure prophylaxis (PrEP) access and use in communities hardest hit by the HIV epidemic persist, further exacerbating ongoing racial/ethnic and socioeconomic disparities in HIV incidence. In these same communities, many patients at risk for HIV seek care for sexually transmitted infections (STIs) in Emergency Departments (EDs), but the structure of traditional ED care is poorly suited to address HIV prevention or provide PrEP. To advance the Prevent objective of the Ending the HIV Epidemic (EHE) initiative, ED2PrEP will leverage an implementation science approach to rigorously test two innovative strategies for increasing PrEP uptake among patients seeking STI care in EDs in one of the 48 EHE-identified geographic hotspots.

DETAILED DESCRIPTION:
Severe inequities in HIV pre-exposure prophylaxis (PrEP) access and use persist among Black and Latinx communities most impacted by the HIV epidemic. The Bronx, NY, with over 90% of the population identifying as Black or Latinx, is an Ending the HIV Epidemic (EHE) priority county with the fifth highest HIV diagnosis rate in the U.S. and the lowest PrEP use in NY. Research on barriers to PrEP engagement indicate that the current structure of PrEP access and management is not consonant with the lives, priorities, or needs of the hardest hit communities, further exacerbating ongoing racial/ethnic and socioeconomic disparities in HIV incidence. Many of the same barriers leading to poor PrEP uptake in Black/Latinx communities also drive members of these communities to seek care for sexually transmitted infections (STIs), a known risk factor for HIV, in Emergency Departments (EDs). However, there is a discordance between the type of care likely to preserve the long-term health of those seeking STI care in EDs (longitudinal, behavioral, and prevention-oriented) and the care the ED is optimized to provide (acute, high intensity, life-saving/stabilizing), meaning that both patients and health systems stand to gain from a restructuring of how STI care is delivered in EDs. Innovative, efficient, and sustainable strategies for identifying and engaging high priority populations for HIV prevention seeking sexual healthcare in EDs are thus needed. The study team therefore proposes ED2PrEP, a pragmatic Type III hybrid effectiveness-implementation trial comparing two different strategies for increasing PrEP uptake among patients at risk for HIV accessing STI care in Bronx EDs. The two strategies are (1) Post-Visit Outreach (PVO) involving proactive outreach to patients following a sexual health-related ED visit. PVO will be initiated by a Sexual Health Navigator who will provide PrEP education, counseling, and linkage to existing sexual health/PrEP clinics. (2) Tele-sexual health (TSH) will involve a real-time telehealth visit with a Sexual Health Provider during sexual health-related ED visits. TSH will also include education, counseling, and linkage, in addition to the provider's ability to prescribe PrEP at the time of the visit. The project will compare the effectiveness of two strategies implemented at two different EDs for 9 months. After the first 9-month study period (Months 1-9), there will be a 1-month wash-out period (Month 10). The study team will then switch the strategies at the two ED study sites for a second 9-month study period (Months 11-19). The trial duration is approximately 31 months total which includes the two-arm implementation-effectiveness trial (19 months) and a follow-up period (12 months). Throughout the study period, the study team will collect quantitative and qualitative data to inform implementation outcomes. Patients will receive TSH the same day of their ED visit or PVO within 7 days of their ED visit. All patients 18+ years old presenting to one of the ED study sites with sexual health-related complaints who fulfill eligibility criteria will be included in the two-arm trial. For this pragmatic trial, no individual participant recruitment is needed, as all relevant outcome data and covariates are routinely collected as part of clinical care and will be extracted from the Montefiore EHR using standard extraction procedures and NYC DOHMH HIV Registry. To ensure that both ED sites are equally prepared to implement TSH, the ED site starting with TSH will receive TSH-specific trainings one week prior to the launch of the trial. For the ED site implementing TSH in the second trial period, the study team will practice TSH workflows and procedures with a clinical champion during the one-month wash-out period. Because the PVO strategy involves outreach by an SHN (not a member of ED staff) only after an ED visit is completed with no other involvement from ED staff, no ED-specific trainings are needed for this strategy. The overall study will also include an implementation science study (quantitative and qualitative sub-studies), an economic and cost analysis and seroconversion ascertainment. The trial period will be preceded by a 3-month Optimization Phase to standardize study workflows and procedures.

ELIGIBILITY:
Inclusion Criteria for Two-Arm Trial:

* Patient is >=18 years at time of index ED visit
* Patient presents to one of the Montefiore ED study sites
* The ED provider applies at least one of the pre-selected ICD-10 CM codes to the encounter and manual review by SHN confirms the visit is related to sexual health

Exclusion Criteria for Two-Arm Trial:

* Patient is admitted to the hospital from the ED
* Known HIV-positive status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1416 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
PrEP Uptake | 3 months
  Prescription of any medication to be used as HIV PrEP, captured in the electronic health record.

SECONDARY OUTCOMES:
PrEP Uptake at 6 months | 6 months
  Prescription of any medication to be used as HIV PrEP, captured in the electronic health record.
PrEP Uptake at 12 months | 12 months
  Prescription of any medication to be used as HIV PrEP, captured in the electronic health record.
Linkage to status neutral healthcare | 3 months
  Attending a clinical appointment for sexual healthcare or related to HIV, captured in the electronic health record
Linkage to status neutral healthcare | 12 months
  Attending a clinical appointment for sexual healthcare or related to HIV, captured in the electronic health record
HIV and STI testing | 6 months
  Receipt of tests for HIV and sexually transmitted infections (gonorrhea and chlamydia from any anatomic site, or syphilis) after the emergency department visit, captured in the electronic health record.
PrEP Persistence | 6 months
  Composite data from the electronic health record about having a prescription for PrEP medications and survey responses about current PrEP use.
PrEP Persistence | 12 months
  Composite data from electronic health record about having a prescription for PrEP medications and survey responses about current PrEP use.
HIV Viral RNA levels | 3 months
  Laboratory quantification of circulating HIV virus among individuals diagnosed with HIV in the study.
HIV Viral RNA levels | 12 months
  Laboratory quantification of circulating HIV virus among individuals diagnosed with HIV in the study.
Incident HIV Diagnosis | 18 months
  Diagnosis of HIV based on multiple data sources (electronic health record, surveys) occurring at anytime starting from ED visit through end of study period.

CONTACTS AND LOCATIONS:
Overall Officials: Uriel Felsen, MD, MS, Principal Investigator — Albert Einstein College of Medicine; Viraj V Patel, MD, MPH, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - City University of New York, New York, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
All deidentified participant level data related to study outcomes.
Supporting Information: Study Protocol, Analytic Code
Time Frame: 6 months after publication of primary outcomes for 5 years.
Access Criteria: Appropriate IRB approvals, research plans approved by study MPIs, and data sharing agreements executed.